CLINICAL TRIAL: NCT06951698
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of KarXT for the Treatment of Manic Episodes in Bipolar-I Disorder (BALSAM-1)
Brief Title: A Study to Evaluate the Efficacy and Safety of KarXT for the Treatment of Manic Episodes in Bipolar-I Disorder
Acronym: BALSAM-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN012-0036; 2024-520165-32 (Other: EU CTR); U1111-1316-7438 (Other: WHO)
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Bipolar-I Disorder With Mania or Mania With Mixed Features
Keywords: Bipolar-I; Mania; Mixed
MeSH Terms: conditions — Mania | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental): Flexible dosing
  Interventions: Drug: KarXT
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline; Trospium Chloride
  Arms: KarXT
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT for the treatment of manic episodes in Bipolar-I Disorder

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter, inpatient study in subjects with bipolar disorder experiencing an acute episode of mania or mania with mixed features.

The primary objective of the study is to evaluate the efficacy of KarXT compared to placebo in treating symptoms of mania during a 3-week inpatient period. The duration of the study including screening, the double-blind inpatient treatment period and safety-follow-up is no more than seven weeks.

ELIGIBILITY:
Inclusion Criteria

* Participants must have a primary diagnosis of Bipolar-I disorder established by a comprehensive psychiatric evaluation.
* Participants must be experiencing an acute episode or relapse of mania or mania with mixed features (≤ 3 weeks).
* Participants must require hospitalization for the acute exacerbation or relapse of mania.
* Participants must have all psychotropic medications washed out in no more than 14 days prior to the first dose of the study drug.
* Participants must have a Young Mania Rating Scale (YMRS) score of ≥ 20 at Screening and at Baseline.
* Participants must have a Clinical Global Impressions-Bipolar (CGI-BP) ≥ 4 at Screening and at Baseline.

Exclusion Criteria:

* Participants must not have any primary Diagnostic and Statistical Manual of Mental Disorders (5th Edition, Text Revision) (DSM-5-TR) disorder, other than BP-I with mania or mania with mixed features within 12 months before screening, including BP-I with depression (for previous 3 months only), BP-II disorder, borderline personality disorder, major depressive disorder, and primary psychotic disorder, with the exception of mild anxiety disorders.
* Participants must not have a primary diagnosis of BP-I with rapid cycling (≥ 4 distinct mood episodes in one year).
* Participants must not have a DSM-5-TR diagnosis of moderate to severe substance use disorder (except tobacco use disorder) within the 12 months before screening, or current use as determined by urine toxicology screen or alcohol test.
* Participants must not be at risk for suicidal behavior at screening or the baseline visit as determined by the Investigator's clinical assessment and the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Participants must not have a history of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months.
* Participants must not have a history or high risk of urinary retention, gastric retention, or untreated narrow-angle glaucoma.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Young Mania Rating Scale (YMRS) score | At week 3
  The YMRS comprised of 11 items that assess the severity of manic symptoms. All items are given a severity rating, with 4 items graded from 0 to 8 (irritability, speech, thought content, and disruptive/aggressive behavior), and the remaining 7 items are graded from 0 to 4 points. The highest score obtainable on the YMRS is 60 and the higher the number the greater the number of symptoms and/or the greater their severity.

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impressions-Bipolar (CGI-BP) | At week 3
  The CGI-BP is designed to assess the severity, improvement, and efficacy of treatment in individuals with bipolar disorder. Only section I, illness severity, will be used, which includes three components: mania, depression, and overall bipolar illness. The ratings are on a 7-point scale (1 = normal, not ill; 2 = minimally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = very severely ill)
Occurrence of response based on a ≥ 50% decrease from baseline in YMRS total score | At week 3
Occurrence of response based on CGI-BP change from baseline ≥ 1 | At week 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (63):
- United States (22):
  - Pillar Clinical Research - Bentonville, Bentonville, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Advanced Research Center Inc., Anaheim, California
  - CITrials, Bellflower, California
  - Local Institution - 0014, Cerritos, California
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - NRC Research Institute, Orange, California
  - Local Institution - 0124, New Haven, Connecticut
  - Health Synergy Clinical Research, Boynton Beach, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - Local Institution - 0015, Miami Lakes, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Pillar Clinical Research -Chicago, Chicago, Illinois
  - Richmond Behavioral Associates, Staten Island, New York
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Local Institution - 0029, Irving, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas
- Argentina (4):
  - Local Institution - 0110, ABB, Buenos Aires F.D.
  - Local Institution - 0115, Córdoba
  - Local Institution - 0108, Mendoza
  - Local Institution - 0109, Mendoza
- Australia (2):
  - Ramsay Clinic Northside, St Leonards, New South Wales
  - Ramsay Clinic New Farm, Brisbane, Queensland
- Bulgaria (5):
  - Center for Mental Health Prof. Dr. Ivan Temkov, Burgas
  - Local Institution - 0119, Novi Iskar
  - Local Institution - 0112, Pleven
  - Local Institution - 0120, Sliven
  - Local Institution - 0121, Vratsa
- Hungary (3):
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Local Institution - 0114, Budapest
  - Semmelweis Egyetem, Budapest
- Japan (19):
  - Local Institution - 0082, Kōnan, Aichi-ken
  - Okehazama Hospital, Toyoake, Aichi-ken
  - National Kohnodai Medical Center., Ichikawa, Chiba
  - Local Institution - 0100, Kitakyushu, Fukuoka
  - Obihiro Kosei Hospital, Obihiro, Hokkaido
  - Goryokai Medical Corporation - Goryokai Hospital, Sapporo, Hokkaido
  - Kansai Medical University Medical Center, Moriguchi, Osaka
  - Rainbow and Sea Hospital, Karatsu-shi, Saga-ken
  - Local Institution - 0081, Iruma, Saitama
  - Saitama Konan Hospital, Kumagaya, Saitama
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Narimasu Kosei Hospital, tabashi City, Tokyo
  - Kuramitsu Hospital, Fukuoka
  - Local Institution - 0077, Miyazaki
  - Osaka Metropolitan University Hospital, Osaka
  - Local Institution - 0084, Osaka
  - Showa Medical University Karasuyama Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata Sakuracho Hospital, Yamagata
- Local Institution - 0055, Auckland, New Zealand
- Poland (7):
  - Local Institution - 0095, Poznan, Greater Poland Voivodeship
  - Local Institution - 0107, Warsaw, Masovian Voivodeship
  - Local Institution - 0094, Bialystok, Podlaskie Voivodeship
  - Local Institution - 0111, Gdansk, Pomeranian Voivodeship
  - Local Institution - 0103, Rybnik, Silesian Voivodeship
  - Local Institution - 0102, Sosnowiec, Silesian Voivodeship
  - Local Institution - 0096, Tuszyn, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description.
Access Criteria: See plan description.
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06951698.html